CLINICAL TRIAL: NCT02481583
Title: Tolerability and Pharmacokinetic Comparison of Oral, Intramuscular and Intravenous Administration of Levosulpiride After Single and Multiple Doses in Fasting Healthy Chinese Volunteers
Brief Title: Pharmacokinetic Study of Levosulpiride
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Weiyong Li, vice director of the pharmacy department, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: WHXH-Levosul
Record Dates: First submitted 2015-05-09; First posted 2015-06-25 (Estimated); Last update posted 2015-06-25 (Estimated); Status verified 2015-06

CONDITIONS: Dyspepsia
Keywords: levosulpiride; pharmacokinetics; adverse effects; bioavailability
MeSH Terms: conditions — Dyspepsia | interventions — levosulpiride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- part 1 (Experimental): 12 subjects successively received a single dose of levosulpiride tablets 25, 50, or 100 mg via oral administration and 50-mg of levosulpiride tablets 3 times a day for 7 days.
  Interventions: Drug: Levosulpiride
- part 2 (Experimental): 30 subjects were randomly assigned to 1 of 3 treatment groups (25, 50, or 75 mg) via i.m. administration, the 50-mg group subjects also received levosulpiride by i.v. route and repeated administration by i.m. route (twice a day for 3 days).
  Interventions: Drug: Levosulpiride

INTERVENTIONS:
Drug: Levosulpiride — different formulations of levosulpiride

SUMMARY:
The aim of this study was to characterise the pharmacokinetic properties and assess the safety of different formulations of levosulpiride in healthy Chinese volunteers.

DETAILED DESCRIPTION:
Levosulpiride was administered to 42 healthy male and female (1:1) subjects as tablet (orally) and injection (intramuscularly and intravenously) formulations. Blood samples were collected at regular intervals after single and multiple drug administration. The concentration of levosulpiride in plasma was determined using a validated high performance liquid chromatography-tandem mass spectrometry method. Non-compartmental analysis was performed to estimate pharmacokinetic parameters. The analysis of variance was used to test for linearity and assess the effect of gender on the pharmacokinetic properties of the study drug. Adverse effects were monitored using investigators' questionnaires and subjects' spontaneous reports, vital sign measurements, hematology, clinical chemistry, and electrocardiogram.

ELIGIBILITY:
Inclusion Criteria:

* body mass index between19 and 24 kg/m2
* negative for HIV and hepatitis B
* had no clinical important findings on health tests
* thorax radiography and ECG with no abnormalities
* normal blood pressure values
* heart rate

Exclusion Criteria:

* any drug treatment within 2 weeks before starting the study
* participation in another clinical study within the previous 3 months
* alcoholism and smoking
* pregnancy
* breast-feeding
* hypocalcemia
* blood donation or participation in other clinical trials within 3 months before enrollment in the study
* sitting blood pressure <80/50 mm Hg or >140/100 mm Hg
* A ventricular rate <60 beats/min or >100 beats/min at rest

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2013-03; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Cmax | two days
  Peak concentration
Area under the curve-AUC | two days
  Area under the curve - plasma concentration
Clearance-CL | two days
  Clearance
Apparent volume of distribution-V | two days
  The apparent volume of distribution

SECONDARY OUTCOMES:
Safety (adverse events) | one month
  adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Weiyong Li, Principal Investigator — HUST/Union Hospital

REFERENCES:
- [Derived] Xu M, Zhou Y, Ni Y, He X, Li H, Sattar H, Chen H, Li W. Tolerability and Pharmacokinetic Comparison of Oral, Intramuscular, and Intravenous Administration of Levosulpiride After Single and Multiple Dosing in Healthy Chinese Volunteers. Clin Ther. 2015 Nov 1;37(11):2458-67. doi: 10.1016/j.clinthera.2015.08.024. Epub 2015 Sep 26. PMID 26404395